CLINICAL TRIAL: NCT06680466
Title: A Multicenter, Ramdomized, Double-Blind, Dose-Regimen Finding, Placebo and Active-Controlled Phase Ⅱ Study to Evaluate the Efficacy and Safety of YZJ-4729 in Patients With Moderate to Severe Acute Pain After Abdominal Surgery
Brief Title: A Phase Ⅱ Study to Evaluate the Efficacy and Safety of YZJ-4729 in Patients With Moderate to Severe Acute Pain After Abdominal Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YZJ-4729-2-01
Record Dates: First submitted 2024-11-01; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Intervention Model Description: Multi center, randomized, double-blind, placebo-controlled, and positive drug parallel controls
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment group 1 (Experimental)
  Interventions: Drug: YZJ-4729
- Treatment group 2 (Experimental)
  Interventions: Drug: YZJ-4729
- Treatment group 3 (Experimental)
  Interventions: Drug: YZJ-4729
- Treatment group 4 (Experimental)
  Interventions: Drug: YZJ-4729
- Morphine (Active Comparator)
  Interventions: Drug: morphine
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: YZJ-4729 — Dose Group 1
  Arms: Treatment group 1
Drug: morphine — morphine,
  Arms: Morphine
Drug: placebo — placebo
  Arms: Placebo
Drug: YZJ-4729 — Dose Group 2
  Arms: Treatment group 2
Drug: YZJ-4729 — Dose Group 3
  Arms: Treatment group 3
Drug: YZJ-4729 — Dose Group 4
  Arms: Treatment group 4

SUMMARY:
Primary Objective： To explore the analgesic efficacy of YZJ-4729 compared with placebo in patients with acute postoperative pain following abdominal surgery.

Secondary Objective： To explore the analgesic efficacy and safety of YZJ-4729 compared with placebo and morphine in patients with acute postoperative pain following abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 and ≤75 years at screening.
2. 18.0 kg/m2≤Body mass index (BMI) ≤28.0 kg/m2
3. American Society of Anesthesiologists (ASA) Physical Status Classification System classification Ⅰ or Ⅱ.
4. Scheduled to undergo abdominal surgery, and estimated duration of the surgery is between 1 hour and 6 hours.
5. NRS ≥ 4 within 4 hours after after extubation of the tracheal tube.
6. Able to understand and comply with the study procedures and requirements, and able to provide written informed consent before any study procedure

Exclusion Criteria:

1. Individuals with a known history of allergy to any component of the investigational drug, or with an allergy or contraindication to anesthetic/analgesic drugs used during surgery;
2. Patients with the following conditions or medical histories:

   1. Comorbid with stroke, Parkinson's syndrome, cognitive impairment, or a history of epilepsy (excluding convulsions caused by high fever in childhood),
   2. Patients with craniocerebral injury, increased intracranial pressure, or brain tumors,
   3. History of difficult airway, obstructive sleep apnea syndrome, bronchial asthma, chronic respiratory system diseases, other severe respiratory system diseases, or acute upper respiratory tract infections within 2 weeks;
   4. History of myocardial infarction or angina within 6 months before screening, or history of severe arrhythmias such as Ⅱ or higher degree atrioventricular block, with a history of New York Heart Association (NYHA) heart function classification class II or above;
   5. History of vestibular dysfunction or motion sickness, or dizziness, nausea, dry retching/vomiting within 1 week before screening;
   6. Comorbid with gastrointestinal system motility disorders (such as reflux esophagitis) or known/suspected gastrointestinal obstruction, including paralytic gastrointestinal obstruction;
   7. Randomized blood glucose ≥11.1 mmol/L or glycated hemoglobin ≥9% during the screening period;
   8. Patients with a clear diagnosis of clinical hypothyroidism;
   9. Presence of other acute or chronic pain conditions before surgery or comorbid with other physical pain that could confound the evaluation of postoperative pain.
3. Hypertension that has not received regular antihypertensive treatment or is poorly controlled despite treatment: during the screening period, systolic blood pressure greater than 160 mmHg, or diastolic blood pressure greater than 100 mmHg (excluding abnormalities during the peri-anesthetic period).
4. Patients with a systolic blood pressure less than 90 mmHg during the screening period (excluding abnormalities during the peri-anesthetic period);
5. Peripheral capillary oxygen saturation (SpO2) <92% in a non-oxygen-supplemented state (excluding abnormalities during the peri-anesthetic period) at screening;
6. Clinically significantly abnormal electrocardiogram, including a QT interval corrected for heart rate (Fridericia; QTcF interval) of > 450 milliseconds in males and > 470 milliseconds in females, at screening.
7. Abnormal liver or kidney function at cscreening: (total bilirubin > upper limit of normal [ULN], aspartate aminotransferase [AST] >1.5 × ULN AND alanine aminotransferase [ALT] >1.5 × ULN, or serum creatinine (Cr) level g >1.5 × ULN;
8. Abnormal coagulation function: Prothrombin time (PT) prolonged by more than 3 seconds above the upper limit of normal and/or Activated Partial Thromboplastin Time (APTT) prolonged by more than 10 seconds above the upper limit of normal.
9. Positive for Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibodies (HCV-Ab), Treponema pallidum antibodies (for syphilis), and Human Immunodeficiency Virus antibodies (HIV-Ab).
10. Use of medications that affect postoperative analgesic effects before randomization:

    1. Continuous use of opioid analgesics for more than 10 days for any reason within 3 months before randomization, or use of opioid analgesics within 5 half-lives before randomization (except permitted by the protocol);
    2. Use of the following medications within 5 half-lives before randomization (or, if half-life is unknown, within within 14 days), including but not limited to: ketamine, nonsteroidal anti-inflammatory drugs (NSAIDs, aspirin is allowed for cardiovascular event prevention, but it must have been stably used for at least 30 days before randomization, with a daily dose ≤100mg/day), alpha-2 adrenergic receptor agonists with analgesic/sedative effects (such as dexmedetomidine, clonidine), glucocorticoid drugs (excluding topical use), antiepileptic drugs, anxiolytics, antipsychotics, sedatives, or other medications that may affect pain assessment;
    3. Use of analgesic Chinese herbal medicines or traditional Chinese patent medicines within 7 days before randomization.
11. Use of monoamine oxidase inhibitors (such as phenelzine, tranylcypromine, selegiline, pargyline, methamphetamine, etc.), selective serotonin reuptake inhibitors (SSRIs), selective serotonin and norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, or triptans within 14 days before randomization.
12. Use of moderate to severe inhibitors/inducers of the liver metabolic enzyme CYP3A4 within 14 days before randomization (such as: enzyme inhibitors - amiodarone, atazanavir, ketoconazole, clarithromycin, itraconazole, etc., enzyme inducers - rifampin, phenytoin sodium, phenobarbital, carbamazepine, etc.).
13. Participated in any clinical trial involving medication (excluding vitamins and minerals) within 3 months prior to screening, except those not involving investigational drugs;
14. History of drug abuse, alcohol poisoning/dependence, or drug misuse within 2 years prior to screening, or those with a positive urine drug screen during the screening period;
15. Women who are pregnant or breastfeeding;
16. Individuals who plan to conceive, are unwilling or unable to use effective contraceptive measures from the screening period to 3 months after the last use of the investigational product, or those who plan to donate sperm/eggs or have plans for egg freezing;
17. Subjects deemed unsuitable to participate in this clinical trial by the investigator.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
The time-weighted sum of differences in resting state pain intensity over 24 hours (SPID24) | 24 hours

SECONDARY OUTCOMES:
The proportion of subjects who did not use rescue analgesics within 0 to 24 hours | 0~24 hours
The time-weighted sum of differences in resting state pain intensity over different perioid | 0-24 hours
Participant ' satisfaction score for analgesia treatment | 24 hours
Investigator satisfaction score for analgesia treatment | 24 hours

OTHER OUTCOMES:
The total dose and times of rescue analgesics | 0-24 hours
Time of first use of rescue analgesics for the first time | 0-24 hours
The sum of resting state pain relief score over 24 hours | 6、12、18、24、12~24 hours
The total number of PCA compressions and the number of effective PCA compressions within 0-24 hours | 0-24 hours
Time to pain relief | 0-24 hours
The median time for the first improvement of at least 1 point on the NRS score | 0-24 hours
The time-weighted sum of differences in movement state pain intensity over different perioid | 6、12、18、24、12~24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China